CLINICAL TRIAL: NCT03781271
Title: ElectroMagnetic-guided Interstitial Catheter Navigation for Gynecological brachyTherapy: A Phase I Trial
Brief Title: ElectroMagnetic-guided Interstitial Catheter Navigation for Gynecological brachyTherapy
Acronym: E-MINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Ananth Ravi, Clinical Operations Lead of Brachytherapy, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 143-2018
Record Dates: First submitted 2018-11-26; First posted 2018-12-19 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cervical Cancer
Keywords: Interstitial Brachytherapy; Electromagnetic tracking; Implant quality; Image guidance
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 arms of patients will undergo standard routine brachytherapy treatment. A part of the treatment involves the placement of catheters. For both arms of the study the placement of these catheters will be assisted by an electromagnetic navigation system. The difference between the arms will be that the navigation system will be used at different times in the course of their brachytherapy treatment to eliminate bias. One group will undergo electromagnetic navigation assisted catheter placement during their first fraction of treatment while the second arm will undergo electromagnetic navigation assisted catheter placement during their third fraction of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fraction 1-Addition of EMN (Experimental): During the fraction 1 insertion, the custom MRI-compatible vaginal cylinder will be placed in the patient, and will contain the 6 degree-of-freedom (DOF) sensor. The electromagnetic navigation system and computer will have been setup in the operating room (OR) prior to the procedure and will be used to actively insert up to 25 catheters into the target. The catheters will be inserted using a custom metallic stylet that has a custom 5-DOF sensor embedded in the tip for tracking its position in real-time. The physician may use ultrasound for assistance in target visualization as well. Catheter deflections will be detected and corrected for in real-time by the radiation oncologist as the catheter is inserted into the patient during the procedure, this will occur when the EM system is in use.
  Interventions: Device: Electromagnetic Navigation
- Fraction 3-Addition of EMN (Experimental): For the second group of patients in the trial the same protocol will be followed as in the first group, the only difference will be that the electromagnetic navigation is used during the second implantation procedure immediately preceding fraction 3 as opposed to fraction 1, the time at which it was used for the first group of patients.
  Interventions: Device: Electromagnetic Navigation

INTERVENTIONS:
Device: Electromagnetic Navigation — Electromagnetic navigation is a form of surgical navigation that can be incorporated into the cervical interstitial brachytherapy workflow to improve the current standards of guidance.

SUMMARY:
Phase I study evaluating the feasibility of using electromagnetic navigation (EMN) for the catheter implantation procedure required of cervical brachytherapy. The addition of EMN to the current HDR brachytherapy workflow has the potential to dramatically improve implant quality and efficiency for the gynecological interstitial brachytherapy program. Implant quality has been reported to be an important predictive factor for local control and late toxicity.

DETAILED DESCRIPTION:
Cervical cancer poses a significant local and global health problem. In 2017 over 1,500 Canadian women were predicted to develop cervical cancer, and another 400 were approximated to die from the disease. Cervical cancer rates have steadily decreased in developed nations largely due to regular gynaecological screening and public human papillomavirus vaccination programs; however, the disease accounts for up to 12% of all female cancer diagnoses in developing nations, and poses a disproportionate burden on aboriginal women across Canada. Much work needs to be done to address disparities in care and treatment for cervical cancer, both in Canada and worldwide.

FIGO stage IA - IB1 is considered localized disease and treated primarily with surgery. In contrast to early stage disease, tumours that extend greater than 4 cm and beyond the cervix are considered locally advanced. The standard of care for locally advanced cervical cancer defined as FIGO stages IB2 - IVA is external beam radiation therapy with concurrent chemotherapy followed by brachytherapy.

Brachytherapy is a crucial component of therapeutic management that has been shown to be associated with improved local control. High dose rate brachytherapy involves the treatment of local bulky disease using a remotely loaded Iridium-192 source. Brachytherapy delivery exploits rapid dose fall off, allowing for the central pelvis to receive a very high dose while sparing the bladder, rectum, sigmoid and small bowel. This dose escalation is beyond what is conventionally achievable using external radiation therapy methods. More specifically, image guided adaptive brachytherapy employing intracavitary applicators allows for dose optimization and improves target dose coverage for limited size tumours.

Intracavitary applicators have been shown to be adequate from covering symmetric small tumours less than 30 cc. However, for large or complex asymmetric tumours with/without vaginal involvement they are not sufficient to cover the target while respecting normal tissue tolerances. To compensate for these limitations, improvements in local control have been achieved using a combined interstitial and intracavitary technique for larger tumours. Combined intracavitary - interstitial applicators have been designed to target tumours that are not adequately covered by intracavitary applicators alone. The addition of the interstitial technique involves the insertion of catheters into the tumour enabling higher dose conformity and normal tissue sparing. This combined technique has been shown in large tumours with extensive parametrial involvement as well as in cases with unfavourable topography to be effective. Employing this combined technique, perineal-based interstitial image guided adaptive brachytherapy makes it possible to deliver higher doses to the high risk clinical target volume without increasing dose to the bladder, rectum or sigmoid.

The combined interstitial and intracavitary brachytherapy workflow for locally advanced cervical cancer at the Odette Cancer Centre typically consists of four treatment fractions. The workflow begins with a pre-brachytherapy assessment MRI that is taken before brachytherapy treatment to assist in preplanning of catheter depth and location. At the time of this MRI the patient will have a vaginal cylinder in place. 1-2 weeks after the MRI, the implant and treatment is performed. Prior to the implantation procedure, the patient is given light sedation and a spinal anesthetic, subsequently a vaginal cylinder (Best Medical Systems, Inc, Springfield VA) is inserted into the patient. A perineal template that contains a central opening is fit on the vaginal cylinder. The template is then advanced until it is appositional on the perineum of the patient. Plastic catheters (6F 24 cm) containing metal stylets are inserted through the template and along the grooves of the vaginal cylinder thereby penetrating the perineum and the vagina, respectively. The number, position and depth of the catheters that are used are based on the pre-brachytherapy assessment MRI. After the implantation procedure the template is sutured to the patient and the patient is transferred to an MRI suite where an image of her anatomy is acquired with the catheters and applicators in place. The patient is then sent for a CT scan that is to be used for treatment planning.

Treatment planning involves the registration of the CT and MR datasets. The MR images are used to identify the soft tissue organs at risk and the targets. The CT is used to identify the catheters implanted in the patient. Using the knowledge of where the applicator/catheters are with respect to the targets and organs at risk, a dose distribution is designed to target the cancer while sparing normal tissue. On the same day as the implantation, one treatment fraction is delivered and the patient is admitted overnight. The next day the patient may as a standard of care, depending on the clinical indication undergo one or two additional fractions, separated by at least 6 hours. A week later the same process for the first two fractions will be repeated for the remaining two fractions.

During the insertion of catheters, it has been recognized that they can converge or diverge as they pierce stiff tissues along the implantation path. Without proper image guidance, a template guided interstitial implant could result in an increase in risk of normal tissue complications. Real-time image guidance for catheter insertion is institution dependent, at the Odette Cancer Centre trans-abdominal ultrasound is used for placement of the tandem and more recently the trans-rectal ultrasound has been investigated for catheter placement. Other forms of real-time catheter guidance used at different centres include fluoroscopy, computed tomography (CT), and magnetic resonance imaging (MRI).

The quality of interstitial brachytherapy implants has been reported to be an important predictive factor for local control and late toxicity. The quality of the implant is dependent on the geometry of the catheters, and real time image guidance for interstitial cervical brachytherapy is markedly lacking.

At the Odette Cancer Centre, a four-patient study was conducted to characterize the amount of catheter deflection and angulation during gynaecological high-dose-rate interstitial brachytherapy. Results from this study demonstrated that the mean value of the maximum catheter deflection at the level of the GTV was 9.1 mm +/- 3.2 mm (range 3.0 - 18.4 mm) and can approach as much as 2 cm at the level of the GTV. Although the catheter deflection observed in this study did not result in any significant dosimetric impact the sample size was small and the authors of the study suggested that further investigation into real-time catheter guidance may be necessary into alleviating this deviation to prevent suboptimal plan quality.

Electromagnetic tracking can minimize the uncertainties related to implant quality. The operation of an electromagnetic tracking device depends on a field generator producing a magnetic field that extends across the anatomy of interest. The tracked sensor in this system induces a distance-dependent voltage that is used to determine the spatial position of the sensor within the volume of interest. This technology is extensively used in clinical practice, examples include, surgical interventions, guidance of biopsies, and motion monitoring.

Electromagnetic navigation can be incorporated into the cervical interstitial brachytherapy workflow as a form of real-time catheter guidance. By incorporating this guidance into the current workflow it is possible that a higher degree of accuracy in catheter placement will be achieved when used in conjunction with image-guided brachytherapy. This study seeks to evaluate the efficacy of electromagnetic navigation on the perineal-based interstitial cervix image-guided brachytherapy workflow as part of a phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with FIGO stage IB2-IVA (locally advanced) cervical cancer being treated with combined 3D interstitial / intracavitary HDR brachytherapy in 4 fractions and concurrent chemotherapy
* Minimum of 2 brachytherapy implantation procedures.
* The Syed-Neblett applicator is indicated for use due to the extent/complexity of the disease
* Given informed consent to take part in the study

Exclusion Criteria:

* Metastatic disease
* Bilateral or unilateral hip prostheses
* Pacemakers

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Plan Target Volume and Organs at Risk Dosimetry | 14 days
  The treatment plans generated during the course of treatment for participants will be evaluated. The evaluation of the treatment plans will use the dose received by specific target structures and the dose received by structures that are defined as organs at risk. The specific metric that will be used represents how much dose is received by a certain percentage of a volume. For example, the D98 GTV refers to how much dose is received by 98 percent of the gross tumour volume. The dose is a value that is measured in the unit, Gray. In addition to the dose constraint for the D98 GTV the other dose constraints that will be used for evaluation purposes are, D90 HR-CTV, D98 HR-CTV, D98 IR-CTV and OAR constraints. A significance level of 5% will be used to identify differences between the dose constraints for treatment plans that are generated when EMN is used and when EMN is not used.

CONTACTS AND LOCATIONS:
Overall Officials: Ananth Ravi, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be made available to relevant stakeholders within the Odette Cancer Centre as these results may assist in the translation of this trial into routine clinical practice.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available within 6 months of study completion.
Access Criteria: Data access requests external to the Odette Cancer Centre will be reviewed by the REB at Sunnybrook Health Science Centre prior to permitting access.